CLINICAL TRIAL: NCT05113082
Title: A Multicentric Observational Retrospective Study on Patients With Short Bowel Syndrome and Chronic Intestinal Failure That Underwent Intestinal Transplantation in Brazil
Brief Title: Retrospective Study on Participants With Short Bowel Syndrome and Chronic Intestinal Failure That Underwent Transplantation in Brazil
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-633-4007
Record Dates: First submitted 2021-11-05; First posted 2021-11-09 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Short Bowel Syndrome (SBS)
Keywords: Chronic Intestinal Failure
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with SBS-IF: Participants with SBS-IF who as part of standard or routine clinical practice, that underwent intestinal transplantation over the last 10 years (both dead and alive at the time of study enrollment) will be observed in this retrospective observational study for 10 months.

SUMMARY:
The main aim of this study is to capture management and treatment outcome data in participants with short bowel syndrome and chronic intestinal failure (SBS-IF) that underwent intestinal transplantation in Brazil.

This study is about collecting data available in the participant's medical record and will also describe the demographic and clinical characteristics of these participants. No medication will be provided to participants in this study.

Clinical data will be collected from a period up to 10 years before the day of the intestinal transplantation. No clinic visits will be required as part of participation in this study.

ELIGIBILITY:
Inclusion Criteria

* Participants with a diagnosis of SBS-IF, who underwent intestinal transplantation between April 2011 to April 2021.
* Participants who have signed the informed consent form (or his/her legal representative). For deceased participants or those with lost to follow-up, an informed consent form (ICF) waiver is acceptable.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with SBS-IF that underwent intestinal transplantation in Brazil.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2022-05-21 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Elapsed Time From the Date of Underlying Condition Diagnosis to the Date of SBS-IF Diagnosis | From start of the study up to end of observation period (up to 10 months)
  Elapsed time from the date of underlying condition diagnosis to the date of SBS-IF diagnosis, according to the information described in the medical records will be presented using a Kaplan-Meier curve. Elapsed time is defined as the amount of time that passes from the beginning of an event to its end.
Elapsed Time From the Date of SBS-IF Diagnosis to the Date of Intestinal Transplant Procedure Indication | From start of the study up to end of observation period (up to 10 months)
  Elapsed time from the date of SBS-IF diagnosis to the date of intestinal transplant procedure indication, according to the information described in the medical records will be presented using a Kaplan-Meier curve. Elapsed time is defined as the amount of time that passes from the beginning of an event to its end.
Elapsed Time From the Date of Intestinal Transplant Indication to the Date of Intestinal Transplant Procedure | From start of the study up to end of observation period (up to 10 months)
  Elapsed time from the date of intestinal transplant indication to the date of intestinal transplant procedure, according to the information described in the medical records will be presented using a Kaplan-Meier curve. Elapsed time is defined as the amount of time that passes from the beginning of an event to its end.

SECONDARY OUTCOMES:
Volume of Parenteral Nutrition and Fluid (Intravenous [IV]) Support From Site Admission Until Intestinal Transplantation During Intestinal Transplantation | From start of the study up to end of observation period (up to 10 months)
  Volume (milliliter/day [mL/day]) of parenteral nutrition and fluid (IV) support from site admission until intestinal transplantation will be summarized using descriptive statistics. Parenteral nutrition is the feeding of nutritional products to a person intravenously, by passing the usual process of eating and digestion.
Number of Participants With Parenteral Nutrition and Fluid (IV) Support From Site Admission Until Intestinal Transplantation | From start of the study up to end of observation period (up to 10 months)
  Number of participants with parenteral nutrition and fluid (IV) support from site admission until intestinal transplantation will be summarized using descriptive statistics. Number of participants with parenteral nutrition and fluid support is calculated by day/week. Parenteral nutrition is the feeding of nutritional products to a person intravenously, by passing the usual process of eating and digestion.
Number of Participants Based on Type of Parenteral Nutrition and Fluid (IV) Support From Site Admission Until Intestinal Transplantation | From start of the study up to end of observation period (up to 10 months)
  Number of Participants based on type (ready to use or individualized) of parenteral nutrition and fluid (IV) support from site admission until intestinal transplantation will be summarized using descriptive statistics. Parenteral nutrition is the feeding of nutritional products to a person intravenously, bypassing the usual process of eating and digestion.
Number of Participants Based on Reasons for Intestinal Transplant Indication | From start of the study up to end of observation period (up to 10 months)
  Number of Participants based on reasons for Intestinal Transplant Indication will be summarized using descriptive statistics.
Number of Participants Based on Each Type of Intestinal Transplant Performed | From start of the study up to end of observation period (up to 10 months)
  Number of participants based on each type of intestinal transplant will be summarized using descriptive statistics.
Number of Participants With Hospitalization Related to SBS-IF Disease Since Site Admission Until Intestinal Transplantation | From start of the study up to end of observation period (up to 10 months)
  Number of participants with hospitalizations per patient per year will be calculated based on the number of hospitalizations during the follow-up period.
Length of Hospitalization Related to SBS-IF Disease | From start of the study up to end of observation period (up to 10 months)
  Length of hospitalization (days) related to SBS-IF disease since site admission until intestinal transplantation will be summarized using descriptive statistics.
Number of Participants With Surgery Performed in SBS-IF Participants | From start of the study up to end of observation period (up to 10 months)
  Number of participants with surgery performed in SBS-IF participants since site admission to intestinal transplantation will be summarized using descriptive statistics.
Number of Participants Based on Reason/Indication for Hospitalization in SBS-IF Participants | From start of the study up to end of observation period (up to 10 months)
  Number of participants based on reason/indication for hospitalization by SBS-IF participants since site admission to intestinal transplantation will be summarized using descriptive statistics.
Percentage of Participants With Each Disease Leading to SBS-IF | From start of the study up to end of observation period (up to 10 months)
  Percentage of participants with each disease/cause leading to SBS-IF will be summarized using descriptive statistics.
Number of Participants Based on Anatomy Site | From start of the study up to end of observation period (up to 10 months)
  Number of participants based on anatomy site will be summarized using descriptive statistics.
Length of the Remaining Bowel | From start of the study up to end of observation period (up to 10 months)
  Length of the remaining bowel will be summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/61bcf2e9f571d4002a64b4b3